CLINICAL TRIAL: NCT04864262
Title: Through the Lens of People With Spinal Cord Injury: Using Photovoice to Prevent Falls
Brief Title: Photovoice for Spinal Cord Injury to Prevent Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kristin Musselman, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-6312
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries
Keywords: Falls; Balance; Photovoice
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photovoice (Experimental)
  Interventions: Other: Photovoice

INTERVENTIONS:
Other: Photovoice — Photovoice is a method that uses photographs and dialogue to share experiences, understand an issue and promote positive change. Group meetings will be held four times throughout the photovoice intervention. The goals of the group meetings are to share knowledge about falls and fall prevention, identify commonalities in the issues raised by the participants, and discuss ways in which these issues could be addressed, both at individual and societal levels. For two photo assignments, participants will be asked to take 4-6 pictures for an assigned question. The question for photo assignment #1 will be 'What decreases your likelihood of falling?' The question for photo assignment #2 will be 'How do you reduce the risk of falling so that you can participate in meaningful activities?' Following each photo assignment, participants will complete an individual semi-structured interview with the peer mentor and the research trainee, who will have a background in physical or occupational therapy.

SUMMARY:
Falls is a health crisis that costs health care systems billions of dollars each year. This crisis is especially relevant for people living with spinal cord injury (SCI) as most of these people will fall at least once per year. Falls can cause injury and a fear of falling, which often causes people to restrict their mobility and daily activities. Despite its importance, fall prevention for people with SCI is understudied, and as a result, there is a lack of treatments to address their high fall risk. We will evaluate a new treatment for fall prevention. Photovoice is a method that uses photographs and dialogue to share experiences, understand an issue and promote positive change. Specifically, we aim to evaluate the effects of photovoice on confidence related to balance and falls, occurrence of falls, participation in daily activities and quality of life among people living with SCI. We also aim to understand participants' experiences with photovoice as a fall prevention program. To achieve these aims, 40 individuals living with SCI will participate in this study. Participants will complete a six-week photovoice program that involves photo assignments, individual interviews and group meetings. The program will be led by a person with SCI and a member of the research team with a background in physical or occupational therapy or kinesiology. Questionnaires will be used throughout the study to measure confidence, participation and quality of life. The occurrence of falls will be tracked for 12 weeks before and after the photovoice program. At the end of the study, each participant's experiences with photovoice will be collected through interviews. The proposed research will address a critical gap in SCI rehabilitation, namely effective fall prevention, to improve well-being after SCI. The research findings will inform the need for, and design of, a larger clinical trial, and has the potential to transform fall prevention after SCI.

The data sharing plan includes sharing study-related information with people living with spinal cord injury. Dissemination activities targeting this group will be developed with input from study participants (e.g., photos may be converted to printed and online art displays and shared through community SCI organizations). Dissemination initiatives will also target health care administrators and rehabilitation clinicians. Study information will be shared with the professional associations representing these groups. To reach researchers in the SCI rehabilitation field, study findings will be presented at academic conferences and in rehabilitation-focused journals.

ELIGIBILITY:
Inclusion Criteria:

1) traumatic or non-traumatic, non-progressive SCI >12 months ago; 2) American Spinal Injury Association Impairment Scale (AIS) rating A-D; 3) ≥18 years old; 4) community-dwelling; 5) experienced >1 fall since sustaining a SCI; 6) free of other conditions besides SCI that affect balance (e.g., vestibular disorder); 7) understand spoken English; and 8) have access and ability to use the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Falls Efficacy Scale - International | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  The 16-item ordinal scale measures how concerned individuals are about falling when they perform both easy and difficult physical and social activities, such as getting dressed/undressed, preparing simple meals, and going out to a social event.
Activities-specific Balance Confidence Scale | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  The ABC Scale asks participants to rate their confidence (from 0% to 100%) in their ability to maintain balance while performing 16 functional tasks in standing or while walking.
Spinal Cord Injury Falls Concern Scale | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  The SCI-FCS is designed to assess falls self-efficacy during daily activities among individuals who are dependent upon a wheelchair for mobility
Wheelchair Use Confidence Scale v.3 | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  It is a measure of one's confidence in using a wheelchair according to six wheelchair-related topics: wheelchair activities, negotiating the physical environment, knowledge and problem-solving, advocacy, managing emotions and managing social situations.

SECONDARY OUTCOMES:
Tracking falls | For 12 weeks after of the photovoice intervention
  Counting the number of falls experienced by participants
Survey of Activities and Fear of Falling in the Elderly | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  The SAFE is a measures of the impact of fear of falling on restriction of activity.
Impact on Participation and Autonomy Questionnaire | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  The IPA is a measure of participation and autonomy across five subscales: autonomy indoors, autonomy outdoors, family roles, social relations, and paid work and education.
Life Satisfaction Questionnaire 9 | Up to 7.5 months; change from start of Baseline (Phase I) to pre-intervention (Phase II) to post-intervention (Phase III) to end of 12-week follow-up
  The LiSAT-9 Is a self-report measure assessing quality of life.

OTHER OUTCOMES:
Final Interview | At study completion, 7.5 months.
  A semi-structured interview will be conducted to explore participants' perceptions of the photovoice intervention following a qualitative descriptive design.

CONTACTS AND LOCATIONS:
Locations (1):
- KITE-Toronto Rehabilitation Institute, UHN, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD is available upon request to the UHN REB for approval to access research participant data.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Sessford J, Kaiser A, Chan K, Alavinia M, Al-Anizi O, Singh H, Munce S, Musselman KE. Impact of a photovoice intervention on fall-related psychological variables, participation levels and quality of life in chronic spinal cord injury. J Spinal Cord Med. 2025 Dec 18:1-14. doi: 10.1080/10790268.2025.2593079. Online ahead of print. PMID 41412174
- [Derived] Sessford JD, Chan K, Kaiser A, Singh H, Munce S, Alavinia M, Musselman KE. Protocol for a single group, mixed methods study investigating the efficacy of photovoice to improve self-efficacy related to balance and falls for spinal cord injury. BMJ Open. 2022 Dec 8;12(12):e065684. doi: 10.1136/bmjopen-2022-065684. PMID 36600385